CLINICAL TRIAL: NCT07365475
Title: Efficacy and Safety of Intra-Arterial Albumin as Adjunct to Mechanical Thrombectomy in Acute Ischemic Stroke: A Multicenter, Prospective, Open-Label, Endpoint-Blinded, Randomized Controlled Clinical Trial (AMASS2)
Brief Title: Efficacy and Safety of Intra-Arterial Albumin as Adjunct to Mechanical Thrombectomy in Acute Ischemic Stroke
Acronym: AMASS2
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Huanhu Hospital (Other)
Responsible Party: Principal Investigator, Ming Wei, PhD, Tianjin Huanhu Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TJHH_WM_20260111
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Acute Ischemic Stroke From Large Vessel Occlusion
Keywords: acute ischemic stroke; large vessel occlusion; mechanical thrombectomy; albumin; neuroprotection
MeSH Terms: conditions — Ischemic Stroke | interventions — Serum Albumin, Human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: independent imaging core laboratory
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Albumin Group (Experimental): Albumin Group Subjects assigned to the albumin treatment group after achieving successful recanalization (eTICI ≥ 2b) confirmed by DSA post-thrombectomy will receive a 20% human albumin solution at a dose of 0.60 g/kg. The solution will be administered as a constant-rate infusion into the proximal internal carotid artery over 20 minutes. Vital signs and potential infusion-related reactions must be closely monitored throughout the procedure.
  Mechanical thrombectomy must be performed using clinically approved devices. The specific technical approach is to be determined by the neurointerventional physician based on the patient's individual clinical condition.
  Interventions: Drug: 20% human serum albumin
- Control Group (No Intervention): Subjects in the control group who have achieved successful recanalization (eTICI ≥ 2b) as confirmed by DSA following mechanical thrombectomy will not receive the investigational infusion and will undergo standard medical management only.
  The mechanical thrombectomy procedure must be performed using clinically approved devices. The specific technical approach is to be determined at the discretion of the neurointerventional physician based on the patient's clinical condition.

INTERVENTIONS:
Drug: 20% human serum albumin — 20% human albumin solution at a dose of 0.60g/kg will be administered as a constant-rate infusion into the proximal internal carotid artery over 20 minutes.
  Arms: Albumin Group

SUMMARY:
Stroke remains a predominant global public health challenge, ranking as the third leading cause of death and the fourth leading contributor to disability-adjusted life years (DALYs). According to the Global Burden of Disease Study 2021, there are approximately 93.8 million prevalent stroke cases and 11.9 million new cases worldwide. China bears one of the heaviest burdens, with over 2 million new cases annually. Acute ischemic stroke (AIS), caused by acute cerebrovascular occlusion, accounts for 80% of all strokes. Approximately 30% of AIS cases result from large vessel occlusion (LVO), which typically carries a poor prognosis due to the extensive area of infarction . Research indicates that early recanalization significantly improves clinical outcomes. Currently, intravenous thrombolysis (IVT) and mechanical thrombectomy (MT) are the standard treatments for achieving recanalization . For LVO-related AIS, MT has become the preferred clinical approach due to its extended therapeutic window and superior recanalization rates . However, despite successful recanalization in over 70% of patients, nearly 50% fail to achieve functional independence at 90 days, and mortality remains above 15% . Therefore, enhancing long-term functional outcomes in post-MT patients is a critical unmet clinical need. Human albumin is the most abundant protein in plasma. Beyond maintaining colloid osmotic pressure, it also possesses multiple biological effects, including anti-inflammatory, anti-platelet aggregation, antioxidant, and endothelial protective properties. We conducted a Phase I clinical trial (AMASS-1) for patients post-mechanical thrombectomy, administering human albumin via the internal carotid artery. The results showed that intra-arterial infusion of 20% human albumin at a dose of 0.60 g/kg was safe, with no significant differences in serious adverse reactions such as mortality [Albumin group (6.7%) vs Control group (6.7%), P > 0.05] and symptomatic intracranial hemorrhage [Albumin group (6.7%) vs Control group (13.3%), P > 0.05] compared to the control group. In summary, albumin adjunctive therapy demonstrates good safety and potential neuroprotective effects in patients after mechanical thrombectomy. To further systematically evaluate its efficacy and safety, we plan to conduct a Phase II clinical trial of mechanical thrombectomy combined with intra-arterial albumin infusion for acute ischemic stroke. This is a multicenter, prospective, open-label, endpoint-blinded, randomized controlled trial designed to evaluate the efficacy and safety of intra-arterial infusion of 20% human serum albumin combined with mechanical thrombectomy versus mechanical thrombectomy alone in patients with acute ischemic stroke due to anterior circulation large vessel occlusion who have achieved recanalization after mechanical thrombectomy. A total of 306 patients are planned to be enrolled and randomly assigned in a 1:1 ratio using a dynamic minimization method to two groups: the Albumin Group (0.6 g/kg 20% human serum albumin plus Mechanical Thrombectomy) and the Control Group (Mechanical Thrombectomy alone). The primary efficacy objective of this study is to evaluate whether immediate intra-arterial infusion of 20% human albumin (0.6 g/kg) via the internal carotid artery following successful recanalization (eTICI ≥2b) improves clinical outcomes in patients with acute anterior circulation large vessel occlusion stroke, compared with mechanical thrombectomy alone. The study also aims to evaluate the safety and feasibility of immediate intra-arterial infusion of 20% human albumin (0.6 g/kg) via the internal carotid artery in patients with acute anterior circulation large vessel occlusion stroke who have achieved successful recanalization (eTICI ≥2b) following standard mechanical thrombectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Acute anterior circulation large vessel occlusion (including ICA/MCA-M1 tandem occlusion or isolated MCA-M1 occlusion) confirmed by CTA, MRA, or DSA, with successful recanalization (eTICI score ≥2b) confirmed by the final intraoperative DSA following mechanical thrombectomy
* Baseline NIHSS scores ≥ 6
* Non-contrast CT ASPECTS ≥6
* Time from stroke onset (or last known well) to arterial puncture within 24 hours
* Pre-stroke functional independence, defined as a modified Rankin Scale (mRS) score <2
* Written informed consent obtained from the patient or a legally authorized representative

Exclusion Criteria:

* Intracranial hemorrhage confirmed by cranial CT or MRI
* Midline shift with significant mass effect on cranial CT or MRI
* Isolated internal carotid artery (ICA) occlusion
* History of heart failure or severe cardiovascular disease, including but not limited to pulmonary hypertension or pericardial effusion
* Hemodynamically unstable arrhythmia (based on patient self-report or detected prior to infusion)
* Symptoms or electrocardiographic evidence of acute myocardial infarction upon admission
* Acute or chronic renal failure (serum creatinine >2.0 mg/dL
* Severe anemia (hematocrit <32%
* Known hypersensitivity to albumin or blood products
* Pregnancy
* Persistent hypertension (blood pressure ≥180/100mmHg) prior to albumin infusion
* Current participation in other clinical trials
* Life expectancy of less than 3 months
* Concomitant severe pulmonary disease, such as chronic obstructive pulmonary disease, pulmonary fibrosis, pleural effusion, or acute respiratory distress syndrome
* Any other condition that, in the opinion of the investigator, renders the patient unsuitable for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
Distribution of mRS scores at 90 (±14) days post-randomization | at 90 (±14) days post-randomization
  Distribution of mRS scores

SECONDARY OUTCOMES:
Proportion of subjects with a favorable outcome at 90 (±14) days post-randomization (defined as mRS 0-2); | at 90 (±14) days post-randomization
  Proportion of subjects with a favorable outcome, defined as mRS 0-2
Proportion of subjects with functional independence at 90 (±14) days post-randomization (defined as mRS 0-1) | at 90 (±14) days post-randomization
  Proportion of subjects with functional independence, defined as mRS 0-1
Infarct volume at 24 (±6) hours post-randomization (measured via MRI-DWI) | at 24 (±6) hours post-randomization
  Infarct volume, measured via MRI-DWI
Infarct volume growth from baseline to 24 (±6) hours post-randomization | from baseline to 24 (±6) hours post-randomization
  Infarct volume growth
Recanalization rate at 24 (±6) hours post-randomization | at 24 (±6) hours post-randomization
  Recanalization rate
NIHSS score at 24 (±6) hours post-randomization | at 24 (±6) hours post-randomization
  NIHSS score
NIHSS score at 7 (±1) days or at discharge, whichever occurs first | at 7 (±1) days or at discharge, whichever occurs first
  NIHSS score
EQ-5D-5L score at 90 (±14) days post-randomization | at 90 (±14) days post-randomization
  EQ-5D-5L score
Proportion of subjects with a Barthel Index (BI) ≥95 at 90 (±14) days post-randomization | at 90 (±14) days post-randomization
  Proportion of subjects with a Barthel Index (BI)
Distribution of mRS scores at 180 (±30) days and 1 year (±30 days) post-randomization | at 180 (±30) days and 1 year (±30 days) post-randomization
  Distribution of mRS scores
Proportion of subjects with a favorable outcome (mRS 0-2) at 180 (±30) days and 1 year (±30 days) post-randomization | at 180 (±30) days and 1 year (±30 days) post-randomization
  Proportion of subjects with a favorable outcome (mRS 0-2)
EQ-5D-5L score at 180 (±30) days and 1 year (±30 days) post-randomization | at 180 (±30) days and 1 year (±30 days) post-randomization
  EQ-5D-5L score
Proportion of subjects with a Barthel Index (BI) ≥95 at 180 (±30) days and 1 year (±30 days) post-randomization | at 180 (±30) days and 1 year (±30 days) post-randomization
  Proportion of subjects with a Barthel Index (BI) ≥95
All-cause mortality within 90 (±14) days post-randomization | within 90 (±14) days post-randomization
  All-cause mortality
Symptomatic intracranial hemorrhage (sICH) at 24 (±6) hours post-randomization (according to ECASS III criteria) | at 24 (±6) hours post-randomization
  Symptomatic intracranial hemorrhage (sICH) ,according to ECASS III criteria
Serious adverse events (SAEs) within 90 (±14) days post-randomization | within 90 (±14) days post-randomization
  SAEs
Adverse events (AEs) within 90 (±14) days post-randomization | within 90 (±14) days post-randomization
  AEs
Early neurological deterioration (END), defined as an increase in NIHSS score of ≥4 points from baseline at 24 hours post-randomization | from baseline at 24 hours post-randomization
  END, defined as an increase in NIHSS score of ≥4 points from baseline at 24 hours post-randomization
Proportion of subjects with severe disability at 90 (±14) days post-randomization (defined as mRS 4-6) | at 90 (±14) days post-randomization
  Proportion of subjects with severe disability , defined as mRS 4-6
Albumin-related adverse events within 90 (±14) days post-randomization | within 90 (±14) days post-randomization
  Albumin-related adverse events
SAEs and AEs within 180 (±30) days post-randomization | within 180 (±30) days post-randomization
  SAEs and AEs
SAEs and AEs within 1 year (±30 days) post-randomization | within 1 year (±30 days) post-randomization
  SAEs and AEs

OTHER OUTCOMES:
Levels of inflammatory cytokines (IL-1β, TNF-α, IL-6, IL-10) in the blood at 24 (±6) hours post-randomization | at 24 (±6) hours post-randomization
  Levels of inflammatory cytokines (IL-1β, TNF-α, IL-6, IL-10) in the blood
Serum albumin and B-type natriuretic peptide (BNP) levels at 24 (±6) hours post-randomization | at 24 (±6) hours post-randomization
  Serum albumin and B-type natriuretic peptide (BNP) levels
Levels of inflammatory cytokines (IL-1β, TNF-α, IL-6, IL-10) in the blood at 7 (±1) days post-randomization or at discharge (whichever occurs first) | at 7 (±1) days post-randomization or at discharge (whichever occurs first)
  Levels of inflammatory cytokines (IL-1β, TNF-α, IL-6, IL-10) in the blood
Serum albumin and BNP levels at 7 (±1) days post-randomization or at dis charge (whichever occurs first) | at 7 (±1) days post-randomization or at dis charge (whichever occurs first)
  Serum albumin and BNP levels
Net water uptake (NWU) at 24 (±6) hours post-randomization | at 24 (±6) hours post-randomization
  Net water uptake (NWU)
Progression of net water uptake from baseline to 24 (±6) hours post-randomization | from baseline to 24 (±6) hours post-randomization
  Progression of net water uptake
Cerebrospinal fluid (CSF) volume at 24 (±6) hours post-randomization | at 24 (±6) hours post-randomization
  Cerebrospinal fluid (CSF) volume
Change in cerebrospinal fluid volume from baseline to 24 (±6) hours post-randomization | from baseline to 24 (±6) hours post-randomization
  Change in cerebrospinal fluid volume
Analysis of the Index for Connectivity via Perivascular Spaces (ALPS index) at 24 (±6) hours post-randomization | at 24 (±6) hours post-randomization
  Analysis of the Index for Connectivity via Perivascular Spaces (ALPS index)